CLINICAL TRIAL: NCT04114032
Title: Evaluating Perioperative Interventions to Improve Patient outComes (EPIC-2): BNP Evaluation Before Surgery Study
Brief Title: BNP Evaluation Before Surgery Study: an Observational Study of Natriuretic Peptide Levels Prior to Surgery.
Acronym: EPIC-2
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Bruce Biccard, Second Chair, Department of Anaesthesia and Perioperative Medicine, Professor, University of Cape Town
Other Study IDs: EPIC-2:BNP
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Surgery, Cardiovascular
Keywords: High risk surgical patients; Risk stratification; Natriuretic peptide testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High-risk elective surgical patients: The patient population to be studied are elective patients for non-cardiac surgery.
  1. Age ≥ 45 years of age.
  2. Undergoing intermediate or major non-cardiac surgery requiring an overnight stay in hospital.
  3. With at least one of the following criteria:
     1. History of ischaemic heart disease or peripheral vascular disease (coronary equivalent)
     2. History of stroke or transient ischaemic attack
     3. History of congestive cardiac failure
     4. Diabetes currently on an oral hypoglycaemic agent or insulin
     5. Serum creatinine >175 µmol/L (>2.0mg/dl)

SUMMARY:
A prospective, multi-centre, observational study of preoperative natriuretic peptide testing for patients undergoing non-cardiac surgery conducted over four weeks.

DETAILED DESCRIPTION:
Identification of high-risk surgical patients requires risk stratification. Current clinical risk stratification tools, e.g. Revised Cardiac Risk Index (RCRI), only have a moderate ability to identify these patients. International guidelines, like Canadian Cardiovascular Society on perioperative cardiovascular risk assessment, advocate that all patients 45 yrs and older or patients >18y rs who have significant cardiovascular disease and who are coming for intermediate to high-risk surgery, should get natriuretic peptide (NP) testing. This is because raised preoperative B-type natriuretic peptides have a strong association with postoperative cardiac complications according to observational studies and meta-analyses.

However, in these patients with significant cardiovascular disease coming for intermediate to high-risk surgery it is unknown how many patients will actually have raised B-type natriuretic peptides. That is, which group of patients have an even higher risk in this already high-risk group. Natriuretic peptide (NP) testing is also expensive.

Further identification of patients that need NP testing will reduce costs and focus efforts on those patients who really need it.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 45 years of age.
2. Undergoing intermediate or major non-cardiac surgery requiring an overnight stay in hospital.
3. With at least one of the following criteria:

   1. History of ischaemic heart disease or peripheral vascular disease (coronary equivalent)
   2. History of stroke or transient ischaemic attack
   3. History of congestive cardiac failure
   4. Diabetes currently on an oral hypoglycaemic agent or insulin
   5. Serum creatinine >175 µmol/L (>2.0mg/dl)

Exclusion Criteria:

1. Patient refusal to participate.
2. Patients presenting for cardiac and obstetric or emergency surgery.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises all non-cardiac patients 45yrs presenting for elective surgery at Groote Schuur-, Somerset-, Paarl-, Victoria-, Mitchell's Plain-, Worcester-, and George Hospital over a period four weeks.
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Raised natriuretic peptide | preoperative
  Determine the prevalence of abnormal (raised) NP in patients with clinical risk criteria.

SECONDARY OUTCOMES:
Risk prediction | preoperative
  The secondary objective is to develop a risk prediction model for those patients who will need preoperative NP screening.

CONTACTS AND LOCATIONS:
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
Undecided